CLINICAL TRIAL: NCT00928590
Title: A Twelve-Month Open-Label Safety Study of Polyquaternium-Preserved DuoTrav APS Dosed Once Daily in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Safety Study of DuoTrav APS in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-09-032; EudraCT Number 2009-013178-42
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: open-angle glaucoma; ocular hypertension; pseudoexfoliation; pigment dispersion
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Duotrav

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DuoTrav APS (Experimental): Travoprost/Timolol Maleate Fixed Combination solution, 1 drop in the study eye(s) once daily, at 9 AM, for 12 months
  Interventions: Drug: Travoprost/Timolol Maleate Fixed Combination solution

INTERVENTIONS:
Drug: Travoprost/Timolol Maleate Fixed Combination solution
  Other Names: DuoTrav APS; DuoTrav (POLYQUAD-preserved)

SUMMARY:
The purpose of this study is to describe the long-term safety of a fixed combination product containing an alternative preservative, dosed once daily for 12 months, in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign an informed consent document.
* Open-angle glaucoma or ocular hypertension who would benefit from a fixed combination medication, in the opinion of the investigator.
* Stable treatment of an IOP-lowering medication.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pregnant, breastfeeding, or not using adequate birth control.
* Best-corrected visual acuity (BCVA) worse than 55 ETDRS letters.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, Ph.D, Study Director — Alcon Research